CLINICAL TRIAL: NCT05336656
Title: Assessment of Analgesics and Sedatives in Mechanically Ventilated Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Wilkes University (Other)
Responsible Party: Principal Investigator, Scott Bolesta, Pharm.D., BCPS, FCCM, FCCP, Associate Professor, Wilkes University
Other Study IDs: 251
Record Dates: First submitted 2022-04-18; First posted 2022-04-20 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: COVID-19; ARDS; Withdrawal Syndrome; Iatrogenic Disease
Keywords: Opioid Withdrawal; Benzodiazepine Withdrawal; Narcotic Withdrawal; Critically ill
MeSH Terms: conditions — COVID-19; Substance Withdrawal Syndrome; Iatrogenic Disease; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The analgesic and sedation requirements in critically ill patients with COVID-19 have yet to be described. There are various factors that are likely affecting the agents being utilized for analgesia and sedation in these patients with little evidence to guide therapy. In addition, such non-evidence based practice may be leading to an increased incidence of iatrogenic withdrawal. The investigators seek to determine the analgesia and sedation requirements in critically ill patients with COVID-19 and report practice patterns that may be associated with iatrogenic withdrawal in these patients. The contribution of the proposed research will be an understanding of current analgesia and sedation use and weaning in critically ill patients with COVID-19, and practice patterns that may indicate the occurrence of iatrogenic withdrawal.

This contribution will be significant because it will determine how analgesics and sedatives are being utilized in critically ill patients with COVID-19, and how their use may be leading to additional morbidity. Data from this initial trial will help support further research on the actual incidence of iatrogenic withdrawal in this patient population. Together such research will help inform practice patterns and therapy recommendations in advance of the next SARS-related outbreak.

DETAILED DESCRIPTION:
The design for this study will be an international retrospective cohort trial. The investigators plan to recruit multiple sites to participate in the study through the use of professional organization list serves and contacts from an ongoing trial being conducted by the investigators (i.e. ALERT-ICU), as well as direct outreach to colleagues and associates of members of the investigator team. Data collection will be performed retrospectively utilizing the electronic medical record system at each participating institution. All data collection will be performed using REDCap, a secure web-based data collection tool that meets the HIPAA (Health Insurance Portability and Accountability Act of 1996) requirements for protection of patient health information. Data collected will include various site and patient demographic data. The investigators will also collect opioid and sedative doses, durations of therapy, weaning of doses, and withdrawal assessments.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age and older admitted to an adult intensive care unit who require invasive mechanical ventilation will be included if they meet one of the following additional criteria: 1. diagnosed with ARDS on or after January 1, 2019; 2. tested positive for COVID-19 and admitted on or after January 1, 2021. Consecutively admitted patients who meet inclusion criteria will be considered for enrollment.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded: surgical and trauma patients, admitted for cardiac arrest, admitted with a primary acute vascular event (e.g. ACS, stroke, etc.), brain injury and/or cerebral edema (e.g. traumatic brain injury, intracranial hemorrhage, subarachnoid hemorrhage, etc.), admitted for status epilepticus, pregnant, receiving extracorporeal membrane oxygenation support.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators anticipate involvement of 30 intensive care unit centers within the United States, Canada, Europe, South America, and Middle East. Each site will contribute 10 patients who meet study criteria.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in cumulative analgesia and sedation dose in appropriate units (e.g. mg, micrograms, etc.) | Three months
  The primary outcome will be the difference in cumulative analgesia and sedation dose 72 hours after ICU admission of patients with ARDS compared to patients with COVID-19. The investigators will compare the groups for differences in types of agents utilized, doses (both average and cumulative) and duration. An additional primary outcome will be the differences in analgesia and sedation weaning requirements between patients with ARDS and COVID-19. Specifically, the investigators will evaluate dosing of analgesics and sedatives during weaning and the use of adjuvant agents (e.g. clonidine) and alternate routes of administration (e.g. oral benzodiazepines).

SECONDARY OUTCOMES:
Patterns of analgesia and sedation weaning as determined by a protocol | Three months
  As a secondary outcome the investigators will evaluate patterns of analgesia and sedative weaning that may indicate the occurrence of withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Marc M Perreault, MSc, PharmD, BCPS, FSCPH, FOPQ, Study Director — Université de Montréal; Lisa Burry, PharmD, FCCP, FCCM, PhD, Study Director — MOUNT SINAI HOSPITAL; Céline Gélinas, RN, PhD, Study Director — Ingram School of Nursing; Kathryn E Smith, PharmD, BCPS, BCCCP, Study Director — Maine Health; Nash Wenner, Student, Study Chair — Wilkes University; Jaycee Blair, Student, Study Chair — Wilkes University; Faizan Ali, Student, Study Chair — Wilkes University
Locations (1):
- Wilkes University, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to share individual participant data specific to each institution through data access groups in RedCap
Supporting Information: Study Protocol, SAP
Time Frame: Twelve months after data collection completed
Access Criteria: Individual site data will be accessible to each specific participating study site.
  Only site investigators will have access to their study site data.

REFERENCES:
- [Result] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Result] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Result] Hanidziar D, Bittner EA. Sedation of Mechanically Ventilated COVID-19 Patients: Challenges and Special Considerations. Anesth Analg. 2020 Jul;131(1):e40-e41. doi: 10.1213/ANE.0000000000004887. No abstract available. PMID 32392023
- [Result] Kahn JM, Andersson L, Karir V, Polissar NL, Neff MJ, Rubenfeld GD. Low tidal volume ventilation does not increase sedation use in patients with acute lung injury. Crit Care Med. 2005 Apr;33(4):766-71. doi: 10.1097/01.ccm.0000157786.41506.24. PMID 15818103
- [Result] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Result] Witenko CJ, Littlefield AJ, Abedian S, An A, Barie PS, Berger K. The Safety of Continuous Infusion Propofol in Mechanically Ventilated Adults With Coronavirus Disease 2019. Ann Pharmacother. 2022 Jan;56(1):5-15. doi: 10.1177/10600280211017315. Epub 2021 May 14. PMID 33985368